CLINICAL TRIAL: NCT02287350
Title: A Phase 4, Open-Label Study of the Pharmacokinetics and Safety of Diclofenac Potassium Oral Solution in Pediatric Subjects (Ages 2-12 Years) With Mild to Moderate Acute Pain
Brief Title: Pharmacokinetics & Safety of Diclofenac Potassium Oral Solution in Ped. Subjects (2-12 Yrs) With Mild-Mod. Acute Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81-0074
Record Dates: First submitted 2014-10-27; First posted 2014-11-10 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Pain
Keywords: pain; moderate pain; mild pain; acute pain; mild acute pain; moderate acute pain; mild or moderate acute pain; NSAID; nonsteroidal anti-inflammatory drug
MeSH Terms: conditions — Pain; Acute Pain; Lymphoma, Follicular | interventions — Diclofenac

ARMS (1):
- diclofenac potassium oral solution (Experimental): 5 mg/mL, liquid form, weight-based dosing, every 6 hours, for up to 4 days.
  Interventions: Drug: diclofenac potassium oral solution

INTERVENTIONS:
Drug: diclofenac potassium oral solution — Administration of diclofenac potassium oral solution, taken by mouth, as needed for mild to moderate acute pain.
  Other Names: diclofenac

SUMMARY:
As part of the Pediatric Research Equity Act (PREA) commitment, the objectives of the study are to characterize the pharmacokinetic (PK) profile and to determine the safety and tolerability of diclofenac potassium oral solution in pediatric subjects experiencing mild to moderate acute pain.

DETAILED DESCRIPTION:
This is an open-label study with pediatric subjects, ages 2-12 years, who will be dosed with diclofenac potassium oral solution, based on weight, every 6 hours as needed for the treatment of mild to moderate acute pain for up to 4 days. PK samples will be collected through 6 hours after the first dose. Safety data will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 2-12 years of age.
* Subjects must be post-op, having mild or moderate acute pain.

Other inclusions apply.

Exclusion Criteria:

* Subject has a known history of allergic reaction, hypersensitivity to diclofenac, aspirin, acetaminophen, or reaction to the non-active ingredients of the study medication.
* Subject has been taking analgesics for 48-72 hours prior to Screening.
* Subject has a history of any GI event greater than 6 months before Screening.
* Subject is currently receiving any medication that is contraindicated for use concomitantly with diclofenac or acetaminophen.
* Subject is requiring treatment for pre-existing hypertension.

Other exclusions apply.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Sheffield, Alabama
  - Stanford, California
  - City of Saint Peters, Missouri
  - Dallas, Texas
  - Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Diclofenac Potassium Oral Solution: 5 mg/mL, liquid form, weight-based dosing, every 6 hours, for up to 4 days.
  diclofenac potassium oral solution: Dosing was individualized based on the subject's weight (at least 20 lbs). Volume per dose was 1 mL, 2 mL, 3 mL, 4 mL, or 5 mL; amount of diclofenac potassium per dose was 5 mg, 10 mg, 15 mg, 20 mg, or 25 mg, respectively. Administration of diclofenac potassium oral solution was by mouth, as needed for mild to moderate acute pain.
Period: Overall Study
Arm/Group | Diclofenac Potassium Oral Solution
Started | 51
Completed | 48
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.4 (3.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: To Characterize the Pharmacokinetic (PK) Profile of a Single Dose of Diclofenac Potassium Oral Solution, With Weight-based Dosing, in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (1 of 8).
Description: • Cmax: maximum concentration (ng/mL)
Time Frame: 6 hours (pre-dose, 15, 30, and 60 min, and 2, 4, and 6 hrs post-dose)
Population: The PK population included all subjects in the Safety population who have at least 1 time point with quantifiable study drug concentration after dosing.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 19
ng/mL
  Cmax (ng/mL): number analyzed (Participants) | 18
  Cmax (ng/mL) | 433.9 (297.53)
  pre-dose concentrations (ng/mL): number analyzed (Participants) | 18
  pre-dose concentrations (ng/mL) | 0.000 (0.0000)
  15 min post-dose concentrations (ng/mL): number analyzed (Participants) | 17
  15 min post-dose concentrations (ng/mL) | 378.471 (315.3756)
  30 min post-dose concentrations (ng/mL) | 260.484 (161.9306)
  60 min post-dose concentrations (ng/mL): number analyzed (Participants) | 18
  60 min post-dose concentrations (ng/mL) | 178.544 (108.9297)
  2 hrs post-dose concentrations (ng/mL): number analyzed (Participants) | 18
  2 hrs post-dose concentrations (ng/mL) | 67.394 (54.5705)
  4 hrs post-dose concentrations (ng/mL): number analyzed (Participants) | 18
  4 hrs post-dose concentrations (ng/mL) | 22.964 (21.4744)
  6 hrs post-dose concentrations (ng/mL): number analyzed (Participants) | 17
  6 hrs post-dose concentrations (ng/mL) | 15.042 (13.0339)

2. Primary Outcome: To Characterize the Pharmacokinetic (PK) Profile of a Single Dose of Diclofenac Potassium Oral Solution, With Weight-based Dosing, in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (2 of 8).
Description: • Tmax: time to maximum concentration (hr)
Time Frame: 6 hours (pre-dose, 15, 30, and 60 min, and 2, 4, and 6 hrs post-dose)
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 18
hr | 0.250 [0.22 to 1.08]

3. Primary Outcome: To Characterize the Pharmacokinetic (PK) Profile of a Single Dose of Diclofenac Potassium Oral Solution, With Weight-based Dosing, in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (3 of 8).
Description: • λz: elimination rate constant (1/hr)
Time Frame: 6 hours (pre-dose, 15, 30, and 60 min, and 2, 4, and 6 hrs post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 17
1/hr | 0.47329 (0.141463)

4. Primary Outcome: To Characterize the Pharmacokinetic (PK) Profile of a Single Dose of Diclofenac Potassium Oral Solution, With Weight-based Dosing, in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (4 of 8).
Description: • t1/2: terminal elimination half-life (hr)
Time Frame: 6 hours (pre-dose, 15, 30, and 60 min, and 2, 4, and 6 hrs post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 17
hr | 1.692 (0.8811)

5. Primary Outcome: To Characterize the Pharmacokinetic (PK) Profile of a Single Dose of Diclofenac Potassium Oral Solution, With Weight-based Dosing, in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (5 of 8).
Description: • AUC 0-t: area under the concentration-time curve from time 0 to last time point (t) where diclofenac could be measured (hr*ng/mL)
Time Frame: 6 hours (pre-dose, 15, 30, and 60 min, and 2, 4, and 6 hrs post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 18
hr*ng/mL | 454.544 (219.3114)

6. Primary Outcome: To Characterize the Pharmacokinetic (PK) Profile of a Single Dose of Diclofenac Potassium Oral Solution, With Weight-based Dosing, in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6 of 8).
Description: • AUC 0-∞: area under the concentration-time curve from time 0 to infinity (∞) (hr*ng/mL)
Time Frame: 6 hours (pre-dose, 15, 30, and 60 min, and 2, 4, and 6 hrs post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 17
hr*ng/mL | 491.915 (244.0359)

7. Primary Outcome: To Characterize the Pharmacokinetic (PK) Profile of a Single Dose of Diclofenac Potassium Oral Solution, With Weight-based Dosing, in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (7 of 8).
Description: • CL/F: apparent clearance (mL/hr).
Time Frame: 6 hours (pre-dose, 15, 30, and 60 min, and 2, 4, and 6 hrs post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 17
mL/hr | 25927.177 (12582.7293)

8. Primary Outcome: To Characterize the Pharmacokinetic (PK) Profile of a Single Dose of Diclofenac Potassium Oral Solution, With Weight-based Dosing, in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (8 of 8).
Description: • Vz/F: apparent volume of distribution (mL).
Time Frame: 6 hours (pre-dose, 15, 30, and 60 min, and 2, 4, and 6 hrs post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 17
mL | 66845.275 (64351.3897)

9. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (1 of 7).
Description: • Treatment emergent AEs (TEAEs)
Time Frame: 4 weeks (first dose of study drug and up to 30 days after the date of the last dose of study drug)
Population: The Safety population included all subjects who have received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
Participants | 16

10. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (2 of 7).
Description: • Serious adverse events (SAEs)
Time Frame: 4 weeks (signed informed consent/assent to 30 days after the last dose of study drug)
Population: The Safety population included all subjects who have received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
Participants | 2

11. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (3 of 7).
Description: • Withdrawals due to AEs
Time Frame: 4 weeks (signed informed consent/assent to 30 days after the last dose of study drug)
Population: The Safety population included all subjects who have received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
Participants | 0

12. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (4 of 7).
Description: • Deaths
Time Frame: 4 weeks (signed informed consent/assent to 30 days after the last dose of study drug)
Population: The Safety population included all subjects who have received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
Participants | 0

13. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (5.1 of 7).
Description: • Changes in vital sign measurements: Temperature (degrees C).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: The Safety population included all subjects who have received at least 1 dose of study drug.
  The data presented are changes from baseline to the final visit. Baseline is defined as the last non-missing measurement taken before first treatment with study drug.
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
degrees C
  Baseline (degrees C) | 36.94 (0.485)
  Final Visit (degrees C): number analyzed (Participants) | 47
  Final Visit (degrees C) | 36.67 (0.492)
  Change from Baseline to Final Visit (degrees C): number analyzed (Participants) | 47
  Change from Baseline to Final Visit (degrees C) | -0.29 (0.511)

14. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (5.2 of 7).
Description: • Changes in vital sign measurements: Pulse Rate (beats/min).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
beats/min
  Baseline (beats/min) | 103.7 (24.41)
  Final Visit (beats/min): number analyzed (Participants) | 47
  Final Visit (beats/min) | 93.4 (16.61)
  Change from Baseline to Final Visit (beats/min): number analyzed (Participants) | 47
  Change from Baseline to Final Visit (beats/min) | -10.5 (17.91)

15. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (5.3 of 7).
Description: • Changes in vital sign measurements: Respiratory Rate (breaths/min).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
breaths/min
  Baseline (breaths/min) | 19.7 (3.55)
  Final Visit (breaths/min): number analyzed (Participants) | 47
  Final Visit (breaths/min) | 19.0 (2.90)
  Change from Baseline to Final Visit (breaths/min): number analyzed (Participants) | 47
  Change from Baseline to Final Visit (breaths/min) | -0.9 (3.93)

16. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (5.4 of 7).
Description: • Changes in vital sign measurements: Systolic Blood Pressure (mmHg).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
mmHg
  Baseline (mmHg) | 110.8 (15.29)
  Final Visit (mmHg): number analyzed (Participants) | 47
  Final Visit (mmHg) | 106.6 (13.08)
  Change from Baseline to Final Visit (mmHg): number analyzed (Participants) | 47
  Change from Baseline to Final Visit (mmHg) | -4.5 (15.45)

17. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (5.5 of 7).
Description: • Changes in vital sign measurements: Diastolic Blood Pressure (mmHg).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
mmHg
  Baseline (mmHg) | 70.1 (12.39)
  Final Visit (mmHg): number analyzed (Participants) | 47
  Final Visit (mmHg) | 65.1 (10.86)
  Change from Baseline to Final Visit (mmHg): number analyzed (Participants) | 47
  Change from Baseline to Final Visit (mmHg) | -5.2 (13.81)

18. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.1 of 7).
Description: • Changes in clinical laboratory results: Hematology - Hematocrit (L/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: The Safety population included all subjects who have received at least 1 dose of study drug.
  The data presented are changes from baseline to the final visit. Baseline is defined as the last measurement taken before first treatment with study drug.
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
L/L
  Baseline (L/L) | 0.357 (0.0264)
  Final Visit (L/L): number analyzed (Participants) | 43
  Final Visit (L/L) | 0.363 (0.0290)
  Change from Baseline to Final Visit (L/L): number analyzed (Participants) | 43
  Change from Baseline to Final Visit (L/L) | 0.006 (0.0269)

19. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.2 of 7).
Description: • Changes in clinical laboratory results: Hematology - Hemoglobin (g/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
g/L
  Baseline (g/L) | 120.5 (10.55)
  Final Visit (g/L): number analyzed (Participants) | 43
  Final Visit (g/L) | 121.0 (10.69)
  Change from Baseline to Final Visit (g/L): number analyzed (Participants) | 43
  Change from Baseline to Final Visit (g/L) | 0.4 (8.20)

20. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.3 of 7).
Description: • Changes in clinical laboratory results: Hematology - Platelet Count (10^9/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
10^9/L
  Baseline (10^9/L) | 315.2 (62.79)
  Final Visit (10^9/L): number analyzed (Participants) | 43
  Final Visit (10^9/L) | 402.2 (109.11)
  Change from Baseline to Final Visit (10^9/L): number analyzed (Participants) | 43
  Change from Baseline to Final Visit (10^9/L) | 85.6 (112.28)

21. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.4 of 7).
Description: • Changes in clinical laboratory results: Hematology - White Blood Cells (10^9/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
10^9/L
  Baseline (10^9/L) | 8.749 (4.7523)
  Final Visit (10^9/L): number analyzed (Participants) | 43
  Final Visit (10^9/L) | 8.807 (2.2423)
  Change from Baseline to Final Visit (10^9/L): number analyzed (Participants) | 43
  Change from Baseline to Final Visit (10^9/L) | -0.054 (4.7766)

22. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.5 of 7).
Description: • Changes in clinical laboratory results: Hematology - Basophils (%).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: % Basophils
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
% Basophils
  Baseline (% Basophils): number analyzed (Participants) | 50
  Baseline (% Basophils) | 0.414 (0.3068)
  Final Visit (% Basophils): number analyzed (Participants) | 42
  Final Visit (% Basophils) | 0.496 (0.3150)
  Change from Baseline to Final Visit (% Basophils): number analyzed (Participants) | 41
  Change from Baseline to Final Visit (% Basophils) | 0.085 (0.2466)

23. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.6 of 7).
Description: • Changes in clinical laboratory results: Hematology - Eosinophils (%).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: % Eosinophils
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
% Eosinophils
  Baseline (% Eosinophils): number analyzed (Participants) | 50
  Baseline (% Eosinophils) | 3.911 (3.2009)
  Final Visit (% Eosinophils): number analyzed (Participants) | 42
  Final Visit (% Eosinophils) | 4.514 (3.1678)
  Change from Baseline to Final Visit(% Eosinophils): number analyzed (Participants) | 41
  Change from Baseline to Final Visit(% Eosinophils) | 0.532 (2.9069)

24. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.7 of 7).
Description: • Changes in clinical laboratory results: Hematology - Neutrophils (%).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: % Neutrophils
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
% Neutrophils
  Baseline (% Neutrophils): number analyzed (Participants) | 50
  Baseline (% Neutrophils) | 49.649 (15.1446)
  Final Visit (% Neutrophils): number analyzed (Participants) | 42
  Final Visit (% Neutrophils) | 48.740 (11.1360)
  Change from Baseline to Final Visit(% Neutrophils): number analyzed (Participants) | 41
  Change from Baseline to Final Visit(% Neutrophils) | -0.791 (17.9732)

25. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.8 of 7).
Description: • Changes in clinical laboratory results: Hematology - Lymphocytes (%).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: % Lymphocytes
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
% Lymphocytes
  Baseline (% Lymphocytes): number analyzed (Participants) | 50
  Baseline (% Lymphocytes) | 37.195 (12.4809)
  Final Visit (% Lymphocytes): number analyzed (Participants) | 42
  Final Visit (% Lymphocytes) | 38.186 (10.4428)
  Change from Baseline to Final Visit(% Lymphocytes): number analyzed (Participants) | 41
  Change from Baseline to Final Visit(% Lymphocytes) | 0.866 (16.2141)

26. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.9 of 7).
Description: • Changes in clinical laboratory results: Hematology - Monocytes (%).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: % Monocytes
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
% Monocytes
  Baseline (% Monocytes): number analyzed (Participants) | 50
  Baseline (% Monocytes) | 8.569 (2.9774)
  Final Visit (% Monocytes): number analyzed (Participants) | 42
  Final Visit (% Monocytes) | 7.859 (2.3952)
  Change from Baseline to Final Visit (% Monocytes): number analyzed (Participants) | 41
  Change from Baseline to Final Visit (% Monocytes) | -0.643 (3.0825)

27. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.10 of 7).
Description: • Changes in clinical laboratory results: Chemistry - Albumin (g/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
g/L
  Baseline (g/L) | 40.882 (4.7314)
  Final Visit (g/L): number analyzed (Participants) | 44
  Final Visit (g/L) | 42.341 (5.2205)
  Change from Baseline to Final Visit (g/L): number analyzed (Participants) | 44
  Change from Baseline to Final Visit (g/L) | 1.114 (3.9131)

28. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.11 of 7).
Description: • Changes in clinical laboratory results: Chemistry - Alkaline Phosphatase (U/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
U/L
  Baseline (U/L) | 219.471 (60.3173)
  Final Visit (U/L): number analyzed (Participants) | 44
  Final Visit (U/L) | 206.545 (54.2160)
  Change from Baseline to Final Visit (U/L): number analyzed (Participants) | 44
  Change from Baseline to Final Visit (U/L) | -10.614 (29.3505)

29. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.12 of 7).
Description: • Changes in clinical laboratory results: Chemistry - ALT (SGPT) (U/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
U/L
  Baseline (U/L) | 21.569 (21.0364)
  Final Visit (U/L): number analyzed (Participants) | 44
  Final Visit (U/L) | 17.727 (11.5383)
  Change from Baseline to Final Visit (U/L): number analyzed (Participants) | 44
  Change from Baseline to Final Visit (U/L) | -1.136 (9.0928)

30. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.13 of 7).
Description: • Changes in clinical laboratory results: Chemistry - AST (SGOT) (U/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
U/L
  Baseline (U/L) | 29.392 (11.4001)
  Final Visit (U/L): number analyzed (Participants) | 44
  Final Visit (U/L) | 25.818 (5.5793)
  Change from Baseline to Final Visit (U/L): number analyzed (Participants) | 44
  Change from Baseline to Final Visit (U/L) | -2.568 (11.1426)

31. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.14 of 7).
Description: • Changes in clinical laboratory results: Chemistry - Bicarbonate (CO2) (mmol/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
mmol/L
  Baseline (mmol/L) | 23.590 (2.1776)
  Final Visit (mmol/L): number analyzed (Participants) | 44
  Final Visit (mmol/L) | 24.748 (2.2748)
  Change from Baseline to Final Visit (mmol/L): number analyzed (Participants) | 44
  Change from Baseline to Final Visit (mmol/L) | 1.109 (2.5307)

32. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.15 of 7).
Description: • Changes in clinical laboratory results: Chemistry - Bilirubin Total (umol/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
umol/L
  Baseline (umol/L) | 4.695 (2.3525)
  Final Visit (umol/L): number analyzed (Participants) | 44
  Final Visit (umol/L) | 4.042 (2.8647)
  Change from Baseline to Final Visit (umol/L): number analyzed (Participants) | 44
  Change from Baseline to Final Visit (umol/L) | -0.319 (3.3429)

33. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.16 of 7).
Description: • Changes in clinical laboratory results: Chemistry - BUN (Urea) (mmol/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
mmol/L
  Baseline (mmol/L) | 4.241 (1.4054)
  Final Visit (mmol/L): number analyzed (Participants) | 44
  Final Visit (mmol/L) | 4.380 (1.4918)
  Change from Baseline to Final Visit (mmol/L): number analyzed (Participants) | 44
  Change from Baseline to Final Visit (mmol/L) | 0.326 (1.4264)

34. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.17 of 7).
Description: • Changes in clinical laboratory results: Chemistry - Chloride (mmol/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
mmol/L
  Baseline (mmol/L) | 102.959 (3.2785)
  Final Visit (mmol/L): number analyzed (Participants) | 44
  Final Visit (mmol/L) | 101.839 (3.1748)
  Change from Baseline to Final Visit (mmol/L): number analyzed (Participants) | 44
  Change from Baseline to Final Visit (mmol/L) | -0.773 (2.7935)

35. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.18 of 7).
Description: • Changes in clinical laboratory results: Chemistry - Creatinine (umol/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
umol/L
  Baseline (umol/L) | 32.032 (13.0954)
  Final Visit (umol/L): number analyzed (Participants) | 44
  Final Visit (umol/L) | 35.260 (12.4928)
  Change from Baseline to Final Visit (umol/L): number analyzed (Participants) | 44
  Change from Baseline to Final Visit (umol/L) | 4.159 (8.3375)

36. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.19 of 7).
Description: • Changes in clinical laboratory results: Chemistry - Glucose (mmol/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
mmol/L
  Baseline (mmol/L): number analyzed (Participants) | 49
  Baseline (mmol/L) | 5.167 (0.7358)
  Final Visit (mmol/L): number analyzed (Participants) | 44
  Final Visit (mmol/L) | 4.851 (0.9318)
  Change from Baseline to Final Visit (mmol/L): number analyzed (Participants) | 42
  Change from Baseline to Final Visit (mmol/L) | -0.361 (0.9477)

37. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.20 of 7).
Description: • Changes in clinical laboratory results: Chemistry - LDH (U/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
U/L
  Baseline (U/L): number analyzed (Participants) | 47
  Baseline (U/L) | 253.085 (75.9762)
  Final Visit (U/L): number analyzed (Participants) | 42
  Final Visit (U/L) | 253.071 (84.4854)
  Change from Baseline to Final Visit (U/L): number analyzed (Participants) | 39
  Change from Baseline to Final Visit (U/L) | -1.256 (100.1911)

38. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.21 of 7).
Description: • Changes in clinical laboratory results: Chemistry - Potassium (mmol/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
mmol/L
  Baseline (mmol/L) | 4.366 (0.4274)
  Final Visit (mmol/L): number analyzed (Participants) | 43
  Final Visit (mmol/L) | 4.337 (0.6764)
  Change from Baseline to Final Visit (mmol/L): number analyzed (Participants) | 43
  Change from Baseline to Final Visit (mmol/L) | -0.038 (0.7428)

39. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.22 of 7).
Description: • Changes in clinical laboratory results: Chemistry - Sodium (mmol/L).
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
mmol/L
  Baseline (mmol/L) | 138.510 (2.7230)
  Final Visit (mmol/L): number analyzed (Participants) | 44
  Final Visit (mmol/L) | 139.818 (2.6787)
  Change from Baseline to Final Visit (mmol/L): number analyzed (Participants) | 44
  Change from Baseline to Final Visit (mmol/L) | 1.409 (2.8228)

40. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.23 of 7).
Description: • Changes in clinical laboratory results: Urinalysis - pH.
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
pH
  Baseline (pH): number analyzed (Participants) | 32
  Baseline (pH) | 6.281 (0.6214)
  Final Visit (pH): number analyzed (Participants) | 41
  Final Visit (pH) | 6.598 (0.8079)
  Change from Baseline to Final Visit (pH): number analyzed (Participants) | 29
  Change from Baseline to Final Visit (pH) | 0.276 (0.8720)

41. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (6.24 of 7).
Description: • Changes in clinical laboratory results: Urinalysis - Specific Gravity.
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Specific Gravity
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
Specific Gravity
  Baseline (Specific Gravity): number analyzed (Participants) | 32
  Baseline (Specific Gravity) | 1.022 (0.0077)
  Final Visit (Specific Gravity): number analyzed (Participants) | 41
  Final Visit (Specific Gravity) | 1.020 (0.0065)
  Change from Baseline to Final Visit (Spec.Gravity): number analyzed (Participants) | 29
  Change from Baseline to Final Visit (Spec.Gravity) | 0.000 (0.0068)

42. Secondary Outcome: To Determine the Safety and Tolerability of Diclofenac Potassium Oral Solution in Pediatric Subjects, Ages 2-12 Years Experiencing Mild to Moderate Acute Pain (7 of 7).
Description: • Physical examination findings including abnormal clinically significant findings
Time Frame: 4 weeks (signed informed consent/assent to the final visit)
Population: The Safety population included all subjects who have received at least 1 dose of study drug.
  The data presented is any new or worsened clinically significant abnormal change from baseline to the final visit. Baseline is defined as the last measurement taken before first treatment with study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Diclofenac Potassium Oral Solution
Number analyzed (Participants) | 51
Participants | 1

ADVERSE EVENTS:
Time Frame: 4 weeks (signed informed consent/assent to 30 days after the last dose of study drug)
Description: The Safety population included all subjects who have received at least 1 dose of study drug.
Arm/Group | Diclofenac Potassium Oral Solution
Serious Adverse Events (participants affected / at risk) | 2/51
Other Adverse Events (participants affected / at risk) | 8/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac Potassium Oral Solution (N=51)
Wound Secretion (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac Potassium Oral Solution (N=51)
Pyrexia (General disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees that sponsor shall have the right to the first publication of the study results which is intended to be a joint, multi-center publication. Following the first publication, the PI may publish study data or results, provided however PI submits the proposed publication to sponsor for review at least 60 days prior to the date of the proposed publication. Sponsor may remove any information that is considered confidential and / or proprietary other than study data.